CLINICAL TRIAL: NCT02260024
Title: A Single Dose Five-way Cross-over Study to Establish an in Vitro/in Vivo Correlation (IVIVC) for Oral Slow Release (SR) Tablets With 0.375 mg Pramipexole in Healthy Male Volunteers
Brief Title: In Vitro/in Vivo Correlation (IVIVC) for Oral Slow Release (SR) Tablets Pramipexole in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 248.560
Record Dates: First submitted 2014-10-07; First posted 2014-10-09 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Healthy

ARMS (6):
- Pramipexole IR (Active Comparator)
  Interventions: Drug: Pramipexole IR tablets
- Pramipexole SR C2 in the fasted state (Experimental)
  Interventions: Drug: Pramipexole SR C2
- Pramipexole SR C2A in the fasted state (Experimental)
  Interventions: Drug: Pramipexole SR C2A
- Pramipexole SR C2B in the fasted state (Experimental)
  Interventions: Drug: Pramipexole SR C2B
- Pramipexole SR C in the fasted state (Experimental)
  Interventions: Drug: Pramipexole SR C
- Pramipexole SR C2 in the fed state (Experimental)
  Interventions: Other: High fat, high caloric meal; Drug: Pramipexole SR C2

INTERVENTIONS:
Other: High fat, high caloric meal
  Arms: Pramipexole SR C2 in the fed state
Drug: Pramipexole IR tablets
  Arms: Pramipexole IR
Drug: Pramipexole SR C
  Arms: Pramipexole SR C in the fasted state
Drug: Pramipexole SR C2
  Arms: Pramipexole SR C2 in the fasted state; Pramipexole SR C2 in the fed state
Drug: Pramipexole SR C2A
  Arms: Pramipexole SR C2A in the fasted state
Drug: Pramipexole SR C2B
  Arms: Pramipexole SR C2B in the fasted state

SUMMARY:
The primary objective of the study was to estimate the magnitude of the error in the prediction of in vivo bioavailability (AUC0-30,Cmax) by means of in vitro dissolution data applying the methods of IVIVC. The secondary objective of the study was to investigate whether the intake of food 30 minutes prior to drug administration affects the systemic exposure of pramipexole SR C2 or not

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects as determined by results of the screening
* Signed written informed consent in accordance with Good Clinical Practice (GCP) and local legislation
* Age ≥ 18 and ≤ 50 years
* BMI ≥ 18.5 and ≤ 29.9 kg/m2

Exclusion Criteria:

* Hypersensitivity to pramipexole or to other dopamine agonists
* Supine systolic blood pressure lower than 110 mmHg and supine diastolic blood pressure lower than 60 mmHg at screening
* Any finding of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24:00 hours) within at least one month or less than ten half-lives of the respective drug before enrolment in the study or during the study
* Use of any drugs which might influence the results of the trial up to 7 days prior to enrolment in the study or during the study
* Participation in another trial with an investigational drug (≤ two months prior to administration or during the trial)
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on in-house trial days
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation (≥ 100 mL within four weeks prior to administration or during the trial)
* Any laboratory value outside the clinically accepted reference range
* Excessive physical activities within the last week before the trial or during the trial

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2005-10; Primary Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
AUC0-30 (area under the concentration time curve of pramipexole in blood plasma over the time interval 0 to 30 h after drug administration) | Up to 30 hours after drug administration
Cmax (maximum measured concentration of pramipexole in blood plasma) | Up to 30 hours after drug administration

SECONDARY OUTCOMES:
AUC0-10 (area under concentration-time curve of pramipexole in blood plasma over the time interval from 0 to the median tmax in the fasted state) | Up to 30 hours after drug administration
AUC0-24 (area under concentration-time curve of pramipexole in blood plasma over the time interval from 0 to 24 h after drug administration), | Up to 24 hours after drug administration
AUC0-∞ (area under the concentration-time curve of pramipexole in blood plasma over the time interval from 0 extrapolated to infinity), | Up to 30 hours after drug administration
tmax (time from dosing to the maximum concentration of pramipexole in blood plasma) | Up to 30 hours after drug administration
λz (terminal rate constant in blood plasma), | Up to 30 hours after drug administration
t½ (terminal half-life of pramipexole in blood plasma) | Up to 30 hours after drug administration
MRTpo (mean residence time of pramipexole in the body after oral administration) | Up to 30 hours after drug administration
CL/F (apparent clearance of pramipexole in the blood plasma after extravascular administration) | Up to 30 hours after drug administration
Vz/F (apparent volume of distribution during the terminal phase (λz) following an extravascular dose) | Up to 30 hours after drug administration
Aet1-t2 (amount of analyte that is eliminated in urine from the time point t1 to time point t2) | Up to 120 hours after drug administration
Number of subjects with adverse events | Up to 7 days after last drug administration
Number of subjects with clinically significant findings in vital signs | Up to 7 days after last drug administration
  pulse rate, blood pressure
Number of subjects with clinically significant findings in laboratory parameters | Up to 7 days after last drug administration
Number of subjects with clinically significant findings in physical examination | Up to 7 days after last drug administration